CLINICAL TRIAL: NCT02818049
Title: Cardiopulmonary Effects of Bronchoalveolar Wash on Patients With Acute Respiratory Distress Syndrome
Acronym: FLOOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patient
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I14033 FLOOD
Record Dates: First submitted 2016-06-15; First posted 2016-06-29 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Bronchioalveolar Lavage
Keywords: Bronchioalveolar Lavage
MeSH Terms: interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bronchoalveolar Lavage (Experimental): BAL was performed in accordance with current practice. Patients are oxygenated with FiO2=1 at least 5 min before the start and 4 h after the procedure. Blood pressure, central venous pressure, heart rate and breathing are monitored by a monitor. O2 saturation (SpO2) is monitored continuously by pulse oximetry.
  Interventions: Procedure: Bronchoalveolar Lavage

INTERVENTIONS:
Procedure: Bronchoalveolar Lavage — BAL was performed in accordance with current practice. Patients are oxygenated with FiO2=1 at least 5 min before the start and 4 h after the procedure. Blood pressure, central venous pressure, heart rate and breathing are monitored by a monitor. O2 saturation (SpO2) is monitored continuously by pulse oximetry.

SUMMARY:
The acute respiratory distress syndrome (ARDS) is a clinical syndrome characterized by an inflammatory pulmonary edema, severe hypoxia and endothelial and epithelial diffuse aggression. A European study estimated that this disease represents 7% of admissions to intensive care. Despite progress on the modalities of mechanical ventilation, mortality is always between 25 and 55%. The definition of this syndrome was recently amended by individualizing three sub groups based on the importance of hypoxemia (mild, moderate and severe). Achieving a bronchoalveolar lavage (BAL) by bronchoscopy remains a gold standard in the initial research of pulmonary infectious cause or secondarily face the suspicion of ventilator-associated pneumonia. Cardio pulmonary consequences of this act are not well known in patients with ARDS. The first studies on the consequences of a bronchoscopy on oxygenation of a patient breathing spontaneously have 40 years. More recent work showed a simple bronchoscopy could in the mechanically ventilated patient cause an average decrease of 26% from the base of PaO2, 10% of the mean arterial pressure (MAP) and a significant increase in cardiac output. The existence of ARDS was an independent risk factor associated with hypoxemia. A study by published in Crit Care Med in 1990 can serve as a reference in ventilated patients benefiting from BAL by bronchoscopy: in a subgroup of 26 patients, 23% of patients required an increase in the fraction of inspired oxygen (FiO2) post procedure. A study compared changes in PaO2/FiO2 after BAL with and without endoscopy among patients without (n = 23) or with pneumonia (n = 11): the decrease in PaO2/FiO2 was significant only in the "pneumonia" group. In a study of 30 patients ventilated but not hypoxic , PaO2 was still reduced by 20% 2 hours after the completion of a BAL in 40% of patients. A retrospective series of 99 ventilated patients but not hypoxic, shows that the BAL was well tolerated in accordance with a pre oxygenation procedure 15 min and by gradually decreasing the FiO 2 after the end of the procedure. BAL also appears well tolerated in a study of 12 patients ventilated under sedation and muscle relaxation, in shock and in need of positive expiratory pressure (PEEP) of at least 10 cm H2O but the authors show a decrease in PaO2 that extends well beyond the end of the intervention. Their conclusion is going to offer less invasive diagnostic techniques for patients with PaO2 less than 60 mm. No study has targeted the respiratory and hemodynamic consequences of this technique depending on the intensity of ARDS (mild, moderate or severe).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients intubated mechanically ventilated
* Patients with ARDS according to the new definition of Berlin
* Patients under sedation / analgesia
* Patients for whom BAL is programmed
* Collection of non-family opposition

Exclusion Criteria:

* PaO2 / FiO2 <50 or any situation which according to investigator would create a risk to the patient during the procedure
* Persistent hypotension despite the administered therapeutic
* Patients tracheotomy
* Patients dying
* Care limitations Patients
* Known allergy to muscle relaxants
* Pregnant woman
* Patients under guardianship or under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
change in PaO2/FiO2 measurement | Baseline and 10 minutes
  Assessment of the change in PaO2/FiO2 in immediate post BAL compared to pre BAL results

CONTACTS AND LOCATIONS:
Overall Officials: VIGNON Philippe, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Limoges University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No